CLINICAL TRIAL: NCT02062437
Title: Multicentric Observational Study Evaluating Clinical and Radiological Results of a Total Hip Arthroplasty Using a Ceramic Friction Pair
Brief Title: Clinical and Radiological Results of Total Hip Arthroplasty Using a Ceramic Friction Pair
Acronym: CERAM
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 1301-T-CERAM-R
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2016-05

CONDITIONS: Hip Replacement; Primary, Secondary or Post-traumatic Osteoarthrosis; Femur Head Necrosis; Congenital Dislocations
Keywords: Arthroplasty; Hip Replacement; Ceramic; Acetabular cup; Femoral stem
MeSH Terms: conditions — Neoplasm Metastasis; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total hip replacement using a ceramic friction pair: Patients treated with total hip replacement using a ceramic friction pair Biolox® Delta, with Meije Duo® stem associated with Dynacup® cup

SUMMARY:
The aim of this study is to assess safety and general performance of total hip arthroplasty, composed of a Meije Duo® femoral stem associated with a Dynacup® cup, and using the friction pair Biolox® Delta Ceramic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient implanted with a primary total hip replacement using a ceramic friction pair including Meije Duo® stem associated with a Dynacup® cup.
* Aged of more than 18 years at the time of the surgery.
* Patient with a follow-up of at least 2 years after surgery based on a consecutive and exhaustive series of patients operated within the inclusion period.
* Able to understand information to participate to the study.

Exclusion Criteria:

* Patient having a tumoral pathology.
* Patient having expressed opposition to the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of European patients with a primary total hip replacement using a ceramic friction pair including Meije Duo® stem associated with a Dynacup® cup.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Piriou, MD, Prof., Principal Investigator — Hôpital Universitaire Raymond Poincaré, Garches - France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients who received the same Total Hip Replacement system for primary hip replacement between July and October 2010 were contacted for study participation.
Groups:
- Total Hip Replacement Using a Ceramic Friction Pair: All patients were treated with a total hip replacement using a ceramic friction pair Biolox® delta, with a Meije Duo® cementless stem with HAP associated with a cementless double coating of plasma sprayed titanium and HAP Dynacup® acetabular cup.
Period: Overall Study
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Started | 132 (132 patients who undergone THR (July-Oct 2010), complying with in/exclusion criteria were identified)
Completed | 80 (80 patients were effectively enrolled, when coming back for their 2-year follow-up visit.)
Not Completed | 52
Not completed — Pt. didn't want to come for the 2y visit | 31
Not completed — Patient not available for the 2y visit | 18
Not completed — Death | 2
Not completed — Pt. couldn't come due to med. condition | 1

BASELINE CHARACTERISTICS:
Population: 132 eligible patients were identified and contacted by the investigators: all patients were still implanted with the same THR system when contacted for study participation, including 2 patients who died before this contact: 80 patients were enrolled and completed the study per protocol at the 2-year follow-up visit without any protocol deviations.
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 42
Region of Enrollment [Number; unit: participants]
  France | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: * Surgical incidents.
  * Post-operative complications.
  * Failure and revisions analysis.
Time Frame: 2-year follow-up visit
Population: The total of 80 patients were seen for their 2-Year follow-up visit.
Measure: Number; unit: participants
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Number analyzed (Participants) | 80
participants | 2

2. Secondary Outcome: General Performance: Mobility
Description: Mobility of the hip is assessed by the maximum value in the range of motions, expressed in degrees (°).
  Normal values (usually observed range of motions) are:
  extension (from 0 to 30°), flexion (from 0 to 120°), abduction (from 0 to 45°), adduction (from 0 to 30°), external rotation (from 0 to 45°) and internal rotation (from 0 to 45°).
  Higher values are the best and a negative value indicates that the patient(s) can't reach the minimum normal range of motion.
Time Frame: Baseline
Population: 80 patients were available but per-protocol some pre-operative data were not available for the analysis of mobilities
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Number analyzed (Participants) | 45
Degrees
  Extension | -1 (6)
  Flexion | 89 (12)
  Adduction | 17 (9)
  Abduction | 20 (10)
  External rotation | 20 (9)
  Internal rotation | 7 (13)

3. Other Pre Specified Outcome: General Performance: Objective Clinical Score (PMA)
Description: Postel Merle d'Aubigne (PMA) rating contains three items; pain, function and hip mobility; each noted 0 to 6 points (0 is the worst possible score and 18 is the best possible PMA score).
Time Frame: Baseline
Population: Within per protocol population, data were not complete to calculate the total PMA score for 3 patients at 2-year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Number analyzed (Participants) | 77
score on a scale
  Pain score | 1.9 (1.1)
  Mobility score | 5.1 (0.9)
  Walking score | 4.5 (0.7)
  Total PMA score | 11.5 (1.7)

4. Secondary Outcome: General Performance: Mobility
Description: as for outcome 2
Time Frame: 2-year Follow-up visit
Population: 80 patients were available but per-protocol some pre-operative data were not available for the analysis of mobilities
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Number analyzed (Participants) | 45
Degrees
  Extension | 0 (1)
  Flexion | 107 (13)
  Adduction | 26 (9)
  Abduction | 34 (9)
  External rotation | 30 (7)
  Internal rotation | 21 (9)

5. Other Pre Specified Outcome: General Performance: Objective Clinical Score (PMA)
Description: as for outcome 3
Time Frame: 2-year follow-up visit
Population: Within per protocol population, data were not complete to calculate the total PMA score for 3 patients at 2-year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Number analyzed (Participants) | 77
score on a scale
  Pain score | 5.8 (0.6)
  Mobility score | 6.0 (1.0)
  Walking score | 5.9 (0.5)
  Total PMA score | 17.7 (1.0)

6. Other Pre Specified Outcome: General Performance: Radiological Assessment.
Description: Radiological assessment is based on :
  * Cup radiological signs of osteolysis or radiolucencies.
  * Stem radiological signs of osteolysis or radiolucencies.
  * Ossifications according to Brooker classification from class I: Ossification around the hip joint. to class IV: shows apparent bone ankylosis of the hip. (i.e Class 0 = no ossification)
  * Other Radiological signs
Time Frame: 2-year Follow-up visit
Population: Patients with X-ray data available
Measure: Number; unit: participants
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Number analyzed (Participants) | 80
participants
  Cups without radiological signs | 80
  Stems without radiological signs | 80
  Ossifications (Brooker classification = 0) | 70
  Ossifications (Brooker classification = 1) | 6
  Ossifications (Brooker classification = 2) | 2
  Ossifications (Brooker classification = 3) | 2
  Ossifications (Brooker classification = 4) | 0
  Other radiological signs | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were collected from surgery to last follow-up visit
Arm/Group | Total Hip Replacement Using a Ceramic Friction Pair
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 1/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Hip Replacement Using a Ceramic Friction Pair (N=80)
Femoral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Spiroid fracture of the thighbone due to patient fall 2 weeks after surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Hip Replacement Using a Ceramic Friction Pair (N=80)
Fracture during surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Partial fracture of the Merckel, no additional procedure has been performed during the surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less